CLINICAL TRIAL: NCT06963047
Title: Ultrasound Use Compared With Standard Care for Diagnosis of Blood Loss After Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Evaluation of Blood Loss After Cesarean Delivery Via US Compared to Standard Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Holy Family Hospital, Nazareth, Israel (Other)
Responsible Party: Principal Investigator, Raed Salim, MD, Head of obstetrics and gynecology departement, Holy Family Hospital, Nazareth, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 309-2025-HFH
Record Dates: First submitted 2025-04-19; First posted 2025-05-08 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Postpartum Period
Keywords: Postpartum anemia; Postpartum hemorrhage; Ultrasound; Cesarean section; Intra-abdominal bleeding
MeSH Terms: conditions — Postpartum Hemorrhage; Hemoperitoneum | interventions — Ultrasonography; Standard of Care

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound group (Active Comparator): Group 1: patients will undergo an abdominal and transvaginal ultrasound examination within 24 hours post-surgery.
  Interventions: Diagnostic Test: Ultrasound
- Standard care group (Active Comparator): Group 2: Candidates will be managed according to the standard care, i.e., without a routine postpartum ultrasound.
  Interventions: Other: Standard care

INTERVENTIONS:
Diagnostic Test: Ultrasound — The purpose of the test is to diagnose and assess the amount of blood loss.
  Arms: Ultrasound group
Other: Standard care — Routine management
  Arms: Standard care group

SUMMARY:
Postpartum hemorrhage and anemia are considered a major health concern due to their impact on maternal morbidity and mortality, quality of life, and maternal cognitive and emotional functioning after delivery, which are particularly important during the critical period of mother-child bonding. Hemoglobin levels in the first 24 hours after delivery do not reflect the lowest point (nadir). The postpartum nadir occurs 48-72 hours after delivery due to the initial redistribution of plasma volume. The aim of this study was to examine whether postpartum ultrasound examination precedes laboratory test results in the diagnosis of anemia due to blood loss after cesarean section.

DETAILED DESCRIPTION:
According to the World Health Organization, postpartum anemia should be recognized as a major health concern, as it affects the quality of life, cognitive and emotional function of the mother, which are particularly important during the critical period of mother-child bonding. Additionally, anemia may impact mother-infant interaction, potentially leading to cognitive delays in infants. Furthermore, postpartum anemia increases the risk of postpartum depression, the need for blood transfusions, length of hospital stays, and hospitalization costs.

Hemoglobin (HB) levels within the first 24 hours postpartum do not reflect the lowest point (nadir). The postpartum nadir occurs 48-72 hours after birth due to initial plasma volume redistribution. Diagnosis is made by measuring HB levels, and anemia is defined when HB is below 10 g at 48 hours postpartum. Postpartum anemia requires immediate treatment upon diagnosis and preferably before discharge.

The incidence of postpartum anemia in developing countries is 50-80%. This high incidence reflects a combination of reasons including under or late diagnosis, lack of awareness, and early hospital discharge.

Postpartum hemorrhage, particularly after cesarean section (CS), is a leading cause of postpartum anemia (HB <10 g%) as well as significant morbidity and mortality. When bleeding occurs into the abdominal cavity, diagnosis is more difficult and delayed, often only detected when vital signs become unstable. Early diagnosis is crucial for proper management of blood loss and life-saving interventions. Diagnosis includes laboratory tests and imaging modalities, and treatment is determined based on severity, ranging from iron supplementation, blood transfusions, and even surgical interventions if necessary.

A certain amount of intra-abdominal fluid is common after most CS. However, there is no standardized reference in gynecological literature regarding what fluid volume is considered normal or pathological after surgery, nor its association with complications such as pain, infection, or prolonged hospitalization. Studies have shown that free intra-abdominal fluid was detected in 73% of patients after CS using CT scans, whereas ultrasound (US) detected fluid in less than 5% of women.

Recently, advanced US technology has become available, including 3D imaging and Doppler technology, which allows for quantitative fluid volume assessment. US is considered a valuable tool for rapid assessment of intra-abdominal free fluid. It is a safe, fast, and non-invasive diagnostic modality that can be used in post-cesarean women to detect and measure intra-abdominal and pelvic fluid, causing minimal patient discomfort. US has several advantages over CT scans and most gynecology departments are equipped with US machines, and gynecologists are trained to use them in clinical practice.

Currently, there is no routine use of US to assess intra-abdominal fluid volume after CS. HB levels are only measured 24 hours post-surgery, which does not necessarily reflect the nadir value. After discharge, many postpartum women may not take iron supplements due to unrecognized anemia, poor tolerance, or low adherence. The aim of this study was to examine whether postpartum ultrasound examination compared to standard care, precedes laboratory test results in the diagnosis of anemia due to blood loss after CS.

ELIGIBILITY:
Inclusion Criteria:

* Women who delivered by a cesarean section.
* Age over 18.
* Fluent in Hebrew or Arabic.
* Signed informed consent form.

Exclusion Criteria:

* Lack of consent or inability to provide informed consent.
* Inability to perform a post-surgical ultrasound, such as post-surgery hospitalization in the intensive care unit.
* Women with preoperative coagulation disorders.
* Women whose clinical condition requires a post-cesarean ultrasound examination.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 276 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin drop of 2g% or more within 24 hours | 24 -72 hours
  The proportion of women with a decrease in Hb levels of over 2 g% identified within 24 hours of surgery in both groups.

SECONDARY OUTCOMES:
HB levels after 48-72 | 72 hours postpartum
  Difference in average HB levels after 48-72 hours between the two study groups
Inferior Vena Cava (IVC) diameter | up to 72 hours postpartum
  Measurement of IVC diameter during inspiration and expiration
IVC collapsibility index | up to 72 hours postpartum
  IVC expiration-IVC inspiration/IVC expiration
Uterine walls diameter | up to 72 hours postpartum
  Measured midway between the fundus and the cervix of the uterus
Uterine endometrial diameter | up to 72 hours postpartum
  Measuring the thickness of the inner layer of the uterus
Uterine length | up to 72 hours postpartum
  Measured from the external cervical os to the fundus
Maximum vertical depth of intra-abdominal fluid | up to 72 hours postpartum
  The measurement will be performed using abdominal and/or vaginal transducer
Urine volume in the bladder | up to 72 hours postpartum
  The measurement will be performed using an abdominal transducer
Rate of women in the study group with intra-abdominal fluid | up to 72 hours postpartum
  The measurement will be performed using abdominal and/or vaginal transducer
Intra-abdominal fluid volume | up to 72 hours postpartum
  The assessment will be performed using abdominal and/or vaginal transducer
Presence of intra-abdominal hematomas | up to 72 hours postpartum
  The assessment will be performed using abdominal and/or vaginal transducer
Objective assessment of intraoperative blood loss | up to 72 hours postpartum
  Calculated blood loss = total blood volume × (prepartum hematocrit - postpartum hematocrit) + total blood volume transfused (if applicable).
Administration of blood products | up to 72 hours postpartum
  Number of blood units administrated
Postoperative fever | up to 72 hours postpartum
  Maternal fever 38C or more
Incidence of women with surgical site infection | Postoperative day 2 to day 7.
  An infection in the part of the body where a surgery took place
Length of hospital stay | up to 10 days postpartum
  Number of days from delivery to discharge
Maternal discomfort during the ultrasound examination | up to 72 hours postpartum
  Measured on a scale of 1 to 5 (1 = no discomfort, 5 = very uncomfortable).

CONTACTS AND LOCATIONS:
Overall Officials: Raed Salim, MD, Study Chair — Holy Family Hospital, Nazareth, Israel
Locations (1):
- Holy family hospital, Nazareth, North, Israel